CLINICAL TRIAL: NCT06905912
Title: Comparison Between FL41 Tinted Spectacles, Biomedics55 Premier Contact Lenses, and Altius Tinted Contact Lenses on Photophobia
Brief Title: Comparison Between Spectacles and Contact Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Dean A. McGee Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17528
Record Dates: First submitted 2024-08-21; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Photophobia
Keywords: Photophobia; Light Sensitivity
MeSH Terms: conditions — Photophobia

STUDY DESIGN:
Masking Description: This trial will not be blinded as the vivid coloration (or lack thereof) of the lens is obvious as to which is worn.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Altius Tinted Contact Lenses (Experimental): Subjects will be asked to wear either of the two tints available for ten days
  Interventions: Device: Biomedics55 Premier contact lenses, and Altius Tinted Contact Lenses

INTERVENTIONS:
Device: Biomedics55 Premier contact lenses, and Altius Tinted Contact Lenses — Biomedics55 Premier contact lenses, and Altius Tinted Contact Lenses

SUMMARY:
Many people suffer from migraine headaches, some more so than others and a common trigger/complaint is light sensitivity, or photophobia1. Some will go to great lengths to avoid light: a dark room with sunglasses on and blankets over the windows, often missing work/school/social activities, etc. Several ocular conditions are accompanied by photophobia, ranging from mild to debilitating.

DETAILED DESCRIPTION:
Burstein et al. describe a shared neuronal pathway between processing light and migraine signals2. Vessels in the dura mater, which are stimulated during migraines, provide input to the Trigeminal Ganglion (TG), which travels to spinal nuclei, which have connections that synapse in the Lateral Posterior Nucleus (LPN). Some intrinsically photosensitive retinal ganglion cells (ipRGC) also synapse through the LPN. The ipRGC are stimulated by light spectra, such as blue light. The crosstalk between the synapses of the ipRGC and pathways from the dura mater vessels causes an overwhelming number of signals that can cause symptoms ranging from cognitive, visual, motor, olfactory, or auditory disfunctions. Thus, it seems reasonable that a reduction in the amount of light stimulation will help alleviate the overload of signals during a migraine, which will decrease the intensity.

FL-41 glasses filter out approximately 50% of blue light and have been shown effective for migraine reduction3. Altius tinted contact lenses filter out 99% of blue light and therefore should be more effective at reducing photophobia. Since the contact lens has direct contact with and coverage of the cornea, no unfiltered stray light is able to enter the eye thus enhancing its efficacy.

ELIGIBILITY:
Two hundred voluntary subjects will be recruited by researching those who have purchased FL-41 tinted spectacles from the Dean McGee Eye Institute Optical Department. If this does not recruit enough subjects then subject referrals will be solicited from the patient population of the Dean McGee Eye Institute and/or neurology clinics throughout the Oklahoma City metro area.

Subjects must meet the following criteria in order to participate in this study:

* Subjects must have worn FL-41 tinted spectacles for at least one month prior to participating in this study.
* Subjects must have at least 20/30 distance visual acuity in each eye while wearing the contact lenses. Altius lenses are currently available in spherical powers from plano to -6.00.
* Subjects must demonstrate the ability to insert and remove contact lenses. Assistance from friends and family is acceptable.
* Subjects must not have an infectious or progressive ocular disease.

Subjects not meeting all of the above criteria will be excluded from participating in this study.

Early Termination:

If a subject feels their photophobia increases to an intolerable level, they can stop wearing that contact lens type and switch to the other the next day or terminate participation in the study. If this occurs, the data from those subjects will still be included in the study data analysis.

If a subject or physician feel that the health of their cornea is at risk, the subject will cease wearing all contact lenses and seek medical care from the Dean McGee Eye Institute.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparing FL-41 Tinted Eyeglasses, Biomedics 55 Premier, and Altius Grey-Green Tinted Contacts | baseline, after 10 days of wearing Biomedics 22 Premier contacts, and after 10 days of wearing Altius colored contacts.
  questionnaires - scale of 1 to 10 - no light sensitivity and 10 extreme light sensitivity

SECONDARY OUTCOMES:
Evaluating FL-41 Tinted Spectacles | immediately after subject finished at least 30 days of wearing the spectacles but before wearing the Biomedics 55 Premier Contacts
  questionnaire - scale 1-10 :1-no light sensitivity and 10 extreme light sensitivity
Evaluating Biomedics 55 Premier Contacts | immediately after subject finished 10 days of wearing the Biomedics 55 premier contact lenses but before wearing the Altius tinted Contacts
  questionnaire - scale 1-10 :1-no light sensitivity and 10 extreme light sensitivity
Evaluating Altius Grey-Green Tinted Contacts | immediately after subject finished 10 days of wearing the grey-green tinted contact lenses
  questionnaire - scale 1-10 :1-no light sensitivity and 10 extreme light sensitivity
Evaluating Altius Amber Tinted Contacts | immediately after subject finished 10 days of wearing the amber tinted contacts
  questionnaire - scale 1-10 :1-no light sensitivity and 10 extreme light sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Dean McGee Eye Institute, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackburn MK, Lamb RD, Digre KB, Smith AG, Warner JE, McClane RW, Nandedkar SD, Langeberg WJ, Holubkov R, Katz BJ. FL-41 tint improves blink frequency, light sensitivity, and functional limitations in patients with benign essential blepharospasm. Ophthalmology. 2009 May;116(5):997-1001. doi: 10.1016/j.ophtha.2008.12.031. PMID 19410958
- [Background] Burstein R, Noseda R, Fulton AB. Neurobiology of Photophobia. J Neuroophthalmol. 2019 Mar;39(1):94-102. doi: 10.1097/WNO.0000000000000766. PMID 30762717
- [Background] Amiri P, Kazeminasab S, Nejadghaderi SA, Mohammadinasab R, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Migraine: A Review on Its History, Global Epidemiology, Risk Factors, and Comorbidities. Front Neurol. 2022 Feb 23;12:800605. doi: 10.3389/fneur.2021.800605. eCollection 2021. PMID 35281991